CLINICAL TRIAL: NCT02352350
Title: The Predictive Value of Prehospital Blood Lactate Measurement Following Out of Hospital Cardiac Arrest (OHCA) and Return of Spontaneous Circulation (ROSC).
Brief Title: Lactate in Cardiac Arrest
Status: Withdrawn | Type: Observational
Why Stopped: Measurement devices unavailable at this time.
Sponsor: University of Florida (Other)
Collaborators: Alachua County Fire Rescue (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201300816
Record Dates: First submitted 2014-12-04; First posted 2015-02-02 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Arrest; Neurological Injury
Keywords: Pre-Hospital Cardiac Arrest; Blood Lactate Level; Neurological Injury
MeSH Terms: conditions — Heart Arrest; Trauma, Nervous System | interventions — cytidylyl-(3'-5')-cytidine; Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Arrest Patients: All adult patients with non traumatic cardiac arrest in Alachua County Florida will have blood lactate levels taken and neurological outcomes performed based on the Cerebral Performance Categories (CPC) Scale
  Interventions: Other: Blood Lactate Levels; Other: Neurological Outcomes

INTERVENTIONS:
Other: Blood Lactate Levels — Blood lactate levels will be performed on all participants.
Other: Neurological Outcomes — Neurological outcomes will be performed on all participants based on the Cerebral Performance Categories (CPC) Scale.
  Other Names: Cerebral Performance Categories (CPC) Scale

SUMMARY:
Blood lactate levels will be measured using a simple handheld device at time of return of spontaneous circulation (ROSC) following out of hospital cardiac arrest (OHCA). Patient outcomes tracked will include rate of survival to hospital discharge, rate of 6 month survival, and neurological status. The hypothesis for this pre-hospital study is to confirm the previous in-hospital findings that very high blood lactate after ROSC is associated with very high mortality and severe neurological impairment.

DETAILED DESCRIPTION:
This will be a prospective observational study of all primary cardiac arrest patients with prehospital (ROSC) in Alachua County, Florida. After Emergency Medical Services (EMS) activation and arrival at scene of a cardiac arrest, paramedics and Emergency Medical Technicians (EMTs) will provide standard Advanced Cardiac Life Support (ACLS) following 2010 guidelines. This may include chest compressions, early identification and shock of ventricular fibrillation and ventricular tachycardia, obtaining intravenous (IV) or intraosseous (IO) access, administration of IV or IO epinephrine, amiodarone, and pressors, oxygenation and ventilation, and other treatments as indicated for reversible causes of cardiac arrest. At time of IV or IO establishment a small blood sample will be obtained the blood will be measured for blood lactate. EMS personnel will be specifically trained to not to delay care or deviate from standard resuscitation protocols to obtain blood lactate sample. Current local paramedic protocols for cardiac arrest and general medical management include obtaining IV access and capillary blood draw and thus blood lactate measurement does not require any additional invasive procedures or medical risk. As medical director of Alachua County Fire Rescue (ACFR) as well as University of Florida faculty member, Dr. Christine Van Dillen oversees paramedic training, protocol development, and quality assurance in Alachua County, Florida. Dr Karl Huesgen is a faculty physician at the University as well, and works closely with ACFR in these regards. These investigators meet regularly with ACFR administration and provide mandatory paramedic and EMT education. Incorporation of lactate measurement into standard cardiac arrest protocols will be accomplished through the monthly administrative updates and monthly in-person training sessions. Adherence to the investigative protocol will be monitored through the standard quality assurance program in which all cardiac arrests are reviewed. Paramedics will have the option of using either capillary or venous blood for lactate measurement. This flexibility is important because cardiac arrests are often chaotic with substantial variability between site of cardiac arrests, timing of return of spontaneous circulation (e.g. if IV access obtained before cardiac rhythm restoration), patient anatomy (e.g. poor venous access), provider resources (e.g. presence of additional rescue personnel), and other factors. Ideally blood lactate measurement will occur at IV insertion, though it may be measured later with equally valid results during fingerstick glucose measurement. Of note, medical providers will be instructed to not perform any additional IV insertions or fingersticks in order to obtain lactate measurements. Patients will be transported as rapidly as possible to local hospitals.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years of age)
* Non-traumatic primary cardiac arrest

Exclusion Criteria:

* Patients with advanced directives precluding resuscitation,
* Traumatic cardiac arrest, and
* Irreversible signs of death (rigor mortis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All primary cardiac arrest patients in Alachua County with prehospital return of spontaneous circulation (ROSC) in Alachua County, FL.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Blood Lactate Levels correlated with survival | Changes in hour 0, approximately hour 12, approximately day 14, and 6 months
Blood Lactate Levels correlated with Neurological Outcomes | Changes in week 2 and 6 months
  Overall Neurologic function will be assessed using available clinical information and Cerebral Performance Categories, a composite measure including available neurologic and clinical assessments CPC 1. Good cerebral performance: conscious, alert, able to work, might have mild neurologic or psychological deficit.
  CPC 2. Moderate cerebral disability: conscious, sufficient cerebral function for independent activities of daily life. Able to work in sheltered environment.
  CPC 3. Severe cerebral disability: conscious, dependent on others for daily support because of impaired brain function. Ranges from ambulatory state to severe dementia or paralysis.
  CPC 4. Coma or vegetative state: any degree of coma without the presence of all brain death criteria. Unawareness, even if appears awake (vegetative state) without interaction with environment; may have spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness.
  CPC 5. Brain death: apnea, areflexia, EEG silence, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Huesgen, MD, Principal Investigator — University of Florida